CLINICAL TRIAL: NCT02392559
Title: Double-blind, Randomized, Multicenter, Placebo-Controlled Study to Characterize the Efficacy, Safety, and Tolerability of 24 Weeks of Evolocumab for LDL-C Reduction in Pediatric Subjects 10 to 17 Years of Age With HeFH
Brief Title: Trial Assessing Efficacy, Safety and Tolerability of Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) Inhibition in Paediatric Subjects With Genetic Low-Density Lipoprotein (LDL) Disorders
Acronym: HAUSER-RCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20120123; 2014-002277-11 (EudraCT Number)
Record Dates: First submitted 2015-02-25; First posted 2015-03-19 (Estimated); Results first posted 2020-07-15 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Heterozygous Familial Hypercholesterolemia
Keywords: Hypercholesterolemia; Elevated Cholesterol; High Cholesterol; Heterozygous Familial Hypercholesterolemia; PCSK9 mutations; Paediatric; pediatric; Childhood Familial Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matching subcutaneous injection every 4 weeks (QM)
  Interventions: Drug: Placebo
- EvoMab 420 mg QM (Experimental): Evolocumab subcutaneous injection QM
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab — Dose of subcutaneous evolocumab every 4 weeks
  Other Names: AMG 145; EvoMab
  Arms: EvoMab 420 mg QM
Drug: Placebo — Dose of subcutaneous placebo treatment every 4 weeks
  Arms: Placebo

SUMMARY:
A study to assess safety and efficacy of evolocumab (AMG-145) in paediatric subjects aged 10-17 years diagnosed with heterozygous familial hypercholesterolemia.

DETAILED DESCRIPTION:
A study to evaluate the effect of 24 weeks of subcutaneous (SC) evolocumab compared with placebo, when added to standard of care, on percent change from baseline in low-density lipoprotein cholesterol (LDL-C) in pediatric subjects 10 to 17 years of age with heterozygous familial hypercholesterolemia (HeFH).

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 10 to ≤ 17 years of age (before 18th birthday)
* Diagnosis of heterozygous familial hypercholesterolemia
* On an approved statin with stable optimized dose for ≥ 4 weeks
* Other lipid-lowering therapy stable for ≥ 4 weeks (fibrates must be stable for ≥ 6 weeks)
* Fasting LDL-C ≥ 130 mg/dL (3.4 mmol/L)
* Fasting triglycerides ≤ 400 mg/dL (4.5 mmol/L)

Exclusion Criteria:

* Type 1 diabetes, or type 2 diabetes that is or poorly controlled
* Uncontrolled hyperthyroidism or hypothyroidism
* Cholesterylester transfer protein (CETP) inhibitor in the last 12 months, or mipomersen or lomitapide in the last 5 months
* Previously received evolocumab or any other investigational therapy to inhibit proprotein convertase subtilisin/kexin type 9 (PCSK9).
* Lipid apheresis within the last 12 weeks prior to screening.
* Homozygous familial hypercholesterolemia

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (63):
- United States (12):
  - Research Site, Farmington, Connecticut
  - Research Site, Wilmington, Delaware
  - Research Site, Iowa City, Iowa
  - Research Site, Towson, Maryland
  - Research Site, Minneapolis, Minnesota
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Salt Lake City, Utah
  - Research Site, Morgantown, West Virginia
- Research Site, Camperdown, New South Wales, Australia
- Austria (3):
  - Research Site, Feldkirch
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Brussels
  - Research Site, La Louvière
  - Research Site, Leuven
- Brazil (4):
  - Research Site, Fortaleza, Ceará
  - Research Site, Vitória, Espírito Santo
  - Research Site, Brasília, Federal District
  - Research Site, São Paulo
- Canada (2):
  - Research Site, Chicoutimi, Quebec
  - Research Site, Québec, Quebec
- Colombia (2):
  - Research Site, Barranquilla, Atlántico
  - Research Site, Floridablanca, Santander Department
- Czechia (3):
  - Research Site, Ostrava-Poruba
  - Research Site, Prague
  - Research Site, Svitavy
- Finland (2):
  - Research Site, Helsinki
  - Research Site, Kuopio
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Research Site, Budapest, Hungary
- Italy (4):
  - Research Site, Palermo
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Torino
- Research Site, Kota Bharu, Kelantan, Malaysia
- Research Site, Amsterdam, Netherlands
- Research Site, Christchurch, New Zealand
- Norway (2):
  - Research Site, Bergen
  - Research Site, Oslo
- Research Site, Gdansk, Poland
- Research Site, Guimarães, Portugal
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Research Site, Ljubljana, Slovenia
- South Africa (2):
  - Research Site, Pretoria, Gauteng
  - Research Site, Parow, Western Cape
- Spain (5):
  - Research Site, Córdoba, Andalusia
  - Research Site, Seville, Andalusia
  - Research Site, Barcelona, Catalonia
  - Research Site, A Coruña, Galicia
  - Research Site, Lugo, Galicia
- Switzerland (2):
  - Research Site, Geneva
  - Research Site, Reinach
- Research Site, Taipei, Taiwan
- Turkey (Türkiye) (2):
  - Research Site, Ankara
  - Research Site, Izmir
- United Kingdom (2):
  - Research Site, Birmingham
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Santos RD, Ruzza A, Hovingh GK, Wiegman A, Mach F, Kurtz CE, Hamer A, Bridges I, Bartuli A, Bergeron J, Szamosi T, Santra S, Stefanutti C, Descamps OS, Greber-Platzer S, Luirink I, Kastelein JJP, Gaudet D; HAUSER-RCT Investigators. Evolocumab in Pediatric Heterozygous Familial Hypercholesterolemia. N Engl J Med. 2020 Oct 1;383(14):1317-1327. doi: 10.1056/NEJMoa2019910. Epub 2020 Aug 29. PMID 32865373
- [Background] Gaudet D, Langslet G, Gidding SS, Luirink IK, Ruzza A, Kurtz C, Lu C, Somaratne R, Raal FJ, Wiegman A. Efficacy, safety, and tolerability of evolocumab in pediatric patients with heterozygous familial hypercholesterolemia: Rationale and design of the HAUSER-RCT study. J Clin Lipidol. 2018 Sep-Oct;12(5):1199-1207. doi: 10.1016/j.jacl.2018.05.007. Epub 2018 May 22. PMID 30318065
- [Background] Gaudet D, Ruzza A, Bridges I, Maruff P, Schembri A, Hamer A, Mach F, Bergeron J, Gaudet I, Pierre JS, Kastelein JJP, Hovingh GK, Wiegman A, Raal FJ, Santos RD. Cognitive function with evolocumab in pediatric heterozygous familial hypercholesterolemia. J Clin Lipidol. 2022 Sep-Oct;16(5):676-684. doi: 10.1016/j.jacl.2022.07.005. Epub 2022 Jul 21. PMID 36210291
- [Derived] Schmidt AF, Carter JL, Pearce LS, Wilkins JT, Overington JP, Hingorani AD, Casas JP. PCSK9 monoclonal antibodies for the primary and secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD011748. doi: 10.1002/14651858.CD011748.pub3. PMID 33078867
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 24 March 2016 to 30 May 2019 at 8 research centers in North America, 30 research centers in Europe, 6 research centers in Latin America, and 3 research centers in Asia Pacific.
Pre-assignment Details: Participants were randomized in a 2:1 ratio to receive 24 weeks of monthly (QM) evolocumab or placebo. Randomization was stratified by screening low-density lipoprotein cholesterol (LDL-C; < 160 mg/dL vs ≥ 160 mg/dL) and age (< 14 years vs ≥ 14 years).
Groups:
- Placebo: Matching subcutaneous injection QM
Period: Overall Study
Arm/Group | Placebo | EvoMab 420 mg QM
Started (Randomized) | 53 | 105
Randomized and Dosed | 53 | 104
Completed | 53 | 104
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: participants who were randomized and dosed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | EvoMab 420 mg QM | Total
Number analyzed (Participants) | 53 | 104 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.7 (2.5) | 13.7 (2.3) | 13.7 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 61 | 88
  Male | 26 | 43 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 46 | 98 | 144
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 2 | 2
  Black (or African American) | 0 | 2 | 2
  White | 44 | 89 | 133
  Other, Not Specified | 9 | 11 | 20
Stratification Factor: Age Group [Number; unit: participants]
  < 14 years | 25 | 48 | 73
  ≥ 14 years | 28 | 56 | 84
Stratification Factor: Screening LDL-C Level [Number; unit: participants]
  < 160 mg/dL | 16 | 33 | 49
  ≥ 160 mg/dL | 37 | 71 | 108
LDL-C [Mean (Standard Deviation); unit: mg/dL] | 183.0 (47.2) | 185.0 (45.0) | 184.3 (45.6)
Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 200.2 (48.2) | 203.8 (47.3) | 202.6 (47.5)
Total Cholesterol/HDL-C Ratio [Mean (Standard Deviation); unit: ratio] | 5.517 (1.492) | 5.702 (1.791) | 5.639 (1.694)
Apolipoprotein B (ApoB) [Mean (Standard Deviation); unit: mg/dL] — Population: participants with a baseline measurement
  mg/dL
    number analyzed (Participants) | 51 | 103 | 154
    (all) | 119.4 (27.9) | 123.3 (27.1) | 122.0 (27.3)
ApoB/Apolipoprotein A1 (ApoA1) Ratio [Mean (Standard Deviation); unit: ratio] — Population: participants with a baseline measurement
  ratio
    number analyzed (Participants) | 51 | 103 | 154
    (all) | 0.938 (0.255) | 0.970 (0.302) | 0.960 (0.287)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 112.0 (12.1) | 110.8 (11.5) | 111.2 (11.7)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 67.2 (8.7) | 66.3 (7.7) | 66.6 (8.1)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 74.3 (11.7) | 74.5 (11.1) | 74.4 (11.2)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 24 in LDL-C
Description: Least squares mean is from the repeated measures model which includes treatment group, stratification factors of age and screening LDL-C (from interactive voice response system [IVRS]), scheduled visit and the interaction of treatment with scheduled visit as covariates. The model uses an unstructured covariance.
Time Frame: Baseline, Week 24
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | EvoMab 420 mg QM
Number analyzed (Participants) | 53 | 104
percent change | -6.23 (3.08) | -44.53 (2.17)
Statistical Analysis 1: Comparison: Placebo vs EvoMab 420 mg QM; Test type: Superiority; p < 0.0001, repeated measures model; treatment difference = -38.30, 95% CI 2-sided [-45.54 to -31.06], Standard Error of Mean 3.66 — Treatment difference uses placebo as the reference
Statistical Analysis 2: Comparison: Placebo vs EvoMab 420 mg QM; Test type: Superiority; p < 0.0001, sequential testing/Hochberg procedure — Adjusted p-value based on a combination of sequential testing and the Hochberg procedure to control the overall significance level for all primary and secondary endpoints; Adjusted p-value is compared to 0.05 to determine statistical significance

2. Secondary Outcome: Mean Percent Change From Baseline to Mean of Weeks 22 and 24 in LDL-C
Description: Least squares mean is from the repeated measures model which includes treatment group, stratification factors of age and screening LDL-C (from IVRS), scheduled visit and the interaction of treatment with scheduled visit as covariates.
Time Frame: Baseline, Week 22, Week 24
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | EvoMab 420 mg QM
Number analyzed (Participants) | 53 | 104
percent change | -5.87 (2.66) | -47.95 (1.92)
Statistical Analysis 1: Comparison: Placebo vs EvoMab 420 mg QM; Test type: Superiority; p < 0.0001, repeated measures model; treatment difference = -42.09, 95% CI 2-sided [-48.34 to -35.83], Standard Error of Mean 3.17 — Treatment difference uses placebo as the reference
Statistical Analysis 2: Comparison: Placebo vs EvoMab 420 mg QM; Test type: Superiority; p < 0.0001, sequential testing/Hochberg procedure — [p-value comment as in outcome 1, analysis 2]; Adjusted p-value is compared to 0.05 to determine statistical significance

3. Secondary Outcome: Change From Baseline to Week 24 in LDL-C
Description: as for outcome 2
Time Frame: Baseline, Week 24
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | EvoMab 420 mg QM
Number analyzed (Participants) | 53 | 104
mg/dL | -9.0 (6.2) | -77.5 (4.4)
Statistical Analysis 1: Comparison: Placebo vs EvoMab 420 mg QM; Test type: Superiority; p < 0.0001, repeated measures model — Treatment difference uses placebo as the reference; treatment difference = -68.6, 95% CI 2-sided [-83.1 to -54.0], Standard Error of Mean 7.3
Statistical Analysis 2: Comparison: Placebo vs EvoMab 420 mg QM; Test type: Superiority; p < 0.0001, sequential testing/Hochberg procedure — [p-value comment as in outcome 1, analysis 2]; Adjusted p-value is compared to 0.05 to determine statistical significance

4. Secondary Outcome: Percent Change From Baseline to Week 24 in Non-HDL-C
Description: as for outcome 2
Time Frame: Baseline, Week 24
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | EvoMab 420 mg QM
Number analyzed (Participants) | 53 | 104
percent change | -6.14 (2.87) | -41.19 (2.01)
Statistical Analysis 1: Comparison: Placebo vs EvoMab 420 mg QM; Test type: Superiority; p < 0.0001, repeated measures model; treatment difference = -35.04, 95% CI 2-sided [-41.79 to -28.30], Standard Error of Mean 3.41 — Treatment difference uses placebo as the reference
Statistical Analysis 2: Comparison: Placebo vs EvoMab 420 mg QM; Test type: Superiority; p < 0.0001, sequential testing/Hochberg procedure — [p-value comment as in outcome 1, analysis 2]; Adjusted p-value is compared to 0.05 to determine statistical significance

5. Secondary Outcome: Percent Change From Baseline to Week 24 in Apoliprotein-B (ApoB)
Description: as for outcome 2
Time Frame: Baseline, Week 24
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | EvoMab 420 mg QM
Number analyzed (Participants) | 53 | 104
percent change | -2.37 (2.70) | -34.85 (1.88)
Statistical Analysis 1: Comparison: Placebo vs EvoMab 420 mg QM; Test type: Superiority; p < 0.0001, repeated measures model; treatment difference = -32.47, 95% CI 2-sided [-38.82 to -26.13], Standard Error of Mean 3.21 — Treatment difference uses placebo as the reference
Statistical Analysis 2: Comparison: Placebo vs EvoMab 420 mg QM; Test type: Superiority; p < 0.0001, sequential testing/Hochberg procedure — [p-value comment as in outcome 1, analysis 2]; Adjusted p-value is compared to 0.05 to determine statistical significance

6. Secondary Outcome: Percent Change From Baseline to Week 24 in Total Cholesterol/HDL-C Ratio
Description: as for outcome 2
Time Frame: Baseline, Week 24
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | EvoMab 420 mg QM
Number analyzed (Participants) | 53 | 104
percent change | -4.66 (2.60) | -34.96 (1.82)
Statistical Analysis 1: Comparison: Placebo vs EvoMab 420 mg QM; Test type: Superiority; p < 0.0001, repeated measures model; treatment difference = -30.30, 95% CI 2-sided [-36.40 to -24.21], Standard Error of Mean 3.09 — Treatment difference uses placebo as the reference
Statistical Analysis 2: Comparison: Placebo vs EvoMab 420 mg QM; Test type: Superiority; p < 0.0001, sequential testing/Hochberg procedure — [p-value comment as in outcome 1, analysis 2]; Adjusted p-value is compared to 0.05 to determine statistical significance

7. Secondary Outcome: Percent Change From Baseline to Week 24 in ApoB:ApoA1 Ratio
Description: as for outcome 2
Time Frame: Baseline, Week 24
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | EvoMab 420 mg QM
Number analyzed (Participants) | 53 | 104
percent change | -0.63 (2.80) | -37.02 (1.95)
Statistical Analysis 1: Comparison: Placebo vs EvoMab 420 mg QM; Test type: Superiority; p < 0.0001, repeated measures model; treatment difference = -36.38, 95% CI 2-sided [-42.97 to -29.80], Standard Error of Mean 3.33 — Treatment difference uses placebo as the reference
Statistical Analysis 2: Comparison: Placebo vs EvoMab 420 mg QM; Test type: Superiority; p < 0.0001, sequential testing/Hochberg procedure — [p-value comment as in outcome 1, analysis 2]; Adjusted p-value is compared to 0.05 to determine statistical significance

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Discontinuation (DC), Fatal TEAEs, and Device-Related TEAEs
Description: An adverse event (AE) is defined as any untoward medical occurrence that does not necessarily have a causal relationship with study treatment. An SAE is defined as an adverse event that: is fatal; is a life threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or other medically important serious event. Events were graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grading scale (1=mild; 2=moderate; 3=severe; 4=life-threatening; 5=death). Events were defined as treatment emergent if they occurred after the first dose of study drug and up to and including 30 days after the last dose or the end of study date, whichever is earlier.
Time Frame: From first dose of study drug up to and including 30 days after the last dose or end of study date (Week 24), whichever was earlier. Mean (SD) duration on study was 5.664 (0.278) and 5.608 (0.137) months for Placebo and EvoMab arms, respectively.
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | EvoMab 420 mg QM
Number analyzed (Participants) | 53 | 104
participants
  All TEAEs | 34 | 64
  Grade ≥ 2 TEAEs | 22 | 46
  Grade ≥ 3 TEAEs | 0 | 4
  Grade ≥ 4 TEAEs | 0 | 0
  Serious TEAEs | 0 | 1
  TEAEs Leading to DC of Study Drug | 0 | 1
  Serious TEAEs Leading to DC of Study Drug | 0 | 0
  Non-Serious TEAEs Leading to DC of Study Drug | 0 | 1
  Fatal TEAEs | 0 | 0
  Device-Related TEAEs | 2 | 3
  Device-Related Grade ≥ 2 TEAEs | 0 | 0
  Device-Related Grade ≥ 3 TEAEs | 0 | 0
  Device-Related Grade ≥ 4 TEAEs | 0 | 0
  Serious Device-Related TEAEs | 0 | 0

9. Secondary Outcome: Number of Participants With Maximum Post-Baseline Laboratory Toxicities of Grade ≥ 3
Description: Laboratory toxicity grading was based on NCI CTCAE grading. Grade 3 indicates severe toxicity and Grade 4 indicates life-threatening toxicity. Values representing a worsening from baseline are shown.
Time Frame: Week 24
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | EvoMab 420 mg QM
Number analyzed (Participants) | 53 | 104
participants
  High Total Bilirubin - Grade 3 | 1 | 0
  High Total Cholesterol - Grade 3 | 1 | 1
  High Uric Acid - Grade 3 | 2 | 8

10. Secondary Outcome: Change From Baseline Over Time in Systolic Blood Pressure
Time Frame: Baseline, Week 4, Week 12, Week 20, Week 22, Week 24
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug. Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | EvoMab 420 mg QM
Number analyzed (Participants) | 53 | 104
mmHg
  Change at Week 4: number analyzed (Participants) | 53 | 103
  Change at Week 4 | -0.1 (11.3) | -0.7 (9.4)
  Change at Week 12 | -0.6 (10.3) | 0.3 (9.6)
  Change at Week 20: number analyzed (Participants) | 50 | 100
  Change at Week 20 | -2.1 (7.7) | 0.1 (10.1)
  Change at Week 22: number analyzed (Participants) | 51 | 101
  Change at Week 22 | 1.0 (10.9) | 1.1 (10.0)
  Change at Week 24: number analyzed (Participants) | 46 | 98
  Change at Week 24 | -0.6 (11.4) | 0.6 (10.7)

11. Secondary Outcome: Change From Baseline Over Time in Diastolic Blood Pressure
Time Frame: Baseline, Week 4, Week 12, Week 20, Week 22, Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | EvoMab 420 mg QM
Number analyzed (Participants) | 53 | 104
mmHg
  Change at Week 4: number analyzed (Participants) | 53 | 103
  Change at Week 4 | -2.5 (9.5) | -1.5 (7.3)
  Change at Week 12 | -2.2 (10.0) | 0.5 (8.9)
  Change at Week 20: number analyzed (Participants) | 50 | 100
  Change at Week 20 | -3.3 (7.6) | -0.6 (7.7)
  Change at Week 22: number analyzed (Participants) | 51 | 101
  Change at Week 22 | -1.5 (9.3) | 2.9 (8.0)
  Change at Week 24: number analyzed (Participants) | 46 | 98
  Change at Week 24 | -0.5 (9.0) | 0.3 (8.6)

12. Secondary Outcome: Change From Baseline Over Time in Heart Rate
Time Frame: Baseline, Week 4, Week 12, Week 20, Week 22, Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | EvoMab 420 mg QM
Number analyzed (Participants) | 53 | 104
beats per minute
  Change at Week 4: number analyzed (Participants) | 53 | 103
  Change at Week 4 | 2.1 (11.0) | 0.1 (10.8)
  Change at Week 12 | -0.5 (11.5) | -1.3 (10.2)
  Change at Week 20: number analyzed (Participants) | 50 | 100
  Change at Week 20 | -1.1 (10.3) | 1.1 (11.5)
  Change at Week 22: number analyzed (Participants) | 51 | 101
  Change at Week 22 | 1.3 (13.5) | -0.6 (11.3)
  Change at Week 24: number analyzed (Participants) | 46 | 98
  Change at Week 24 | 0.2 (13.0) | -1.8 (11.8)

13. Secondary Outcome: Number of Participants Testing Positive for Anti-Evolocumab Antibodies
Time Frame: up to Week 24
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug. Participants receiving evolocumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EvoMab 420 mg QM
Number analyzed (Participants) | 0 | 104
Participants
  Binding antibody positive at anytime |  | 0
  Neutralizing antibody positive at anytime |  | 0

14. Secondary Outcome: Serum Evolocumab Concentrations Over Time
Time Frame: Week 12, Week 22, Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | EvoMab 420 mg QM
Number analyzed (Participants) | 99
ng/mL
  Week 12 | 22400 (14700)
  Week 22: number analyzed (Participants) | 81
  Week 22 | 64900 (34400)
  Week 24: number analyzed (Participants) | 96
  Week 24 | 25800 (19200)

ADVERSE EVENTS:
Time Frame: Fatal AEs: from first dose date to end of study date (Week 24); non-fatal AEs: from first dose of study drug up to 30 days after last dose or end of study date, whichever was earlier. Mean (SD) duration on study was 5.664 (0.278) and 5.608 (0.137) months for the Placebo and EvoMab arms, respectively.
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- Placebo SC QM: Matching subcutaneous injection QM
- EvoMab 420 mg SC QM: Evolocumab subcutaneous injection QM
Arm/Group | Placebo SC QM | EvoMab 420 mg SC QM
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/53 | 1/104
Other Adverse Events (participants affected / at risk) | 19/53 | 41/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo SC QM (N=53) | EvoMab 420 mg SC QM (N=104)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo SC QM (N=53) | EvoMab 420 mg SC QM (N=104)
Constipation (Gastrointestinal disorders) | 0 | 3
Influenza like illness (General disorders) | 0 | 3
Pyrexia (General disorders) | 3 | 3
Gastroenteritis (Infections and infestations) | 4 | 5
Influenza (Infections and infestations) | 2 | 6
Nasopharyngitis (Infections and infestations) | 6 | 12
Rhinitis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 6
Blood creatine phosphokinase increased (Investigations) | 2 | 1
Headache (Nervous system disorders) | 1 | 11
Depression (Psychiatric disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2015-09-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT02392559/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT02392559/SAP_001.pdf